CLINICAL TRIAL: NCT00386698
Title: Evaluate Reactogenicity & Immunogenicity of Adjuvanted Influenza Vaccine in Elderly Adults Previously Vaccinated With the Same Candidate Vaccine. Fluarix™ Administered in Young & Elderly Adults Will be Used as Reference
Brief Title: Study to Evaluate Reactogenicity and Immunogenicity of Revaccination With Adjuvanted Influenza Vaccine in Elderly Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 104887
Record Dates: First submitted 2006-10-09; First posted 2006-10-11 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-10

CONDITIONS: Influenza
Keywords: Influenza,; improved vaccine,; influenza disease; elderly
MeSH Terms: conditions — Influenza, Human | interventions — fluarix

INTERVENTIONS:
Biological: Fluarix
Biological: adjuvanted influenza vaccine

SUMMARY:
Since influenza vaccines are normally administered every year because of the frequent change in their antigenic composition, the safety and immunogenicity profiles of the adjuvanted influenza vaccine need to be re-evaluated after repeated vaccine administration. In this study, subjects enrolled in a previous study will receive a booster dose with the 2006-2007 season's formulations of Fluarix or the adjuvanted vaccine.

ELIGIBILITY:
Inclusion Criteria:

* The subjects must be healthy adults ages 18-40 years or >/= 65 years previously vaccinated with either Fluarix or the adjuvanted vaccine.

Exclusion Criteria:

* Subjects will be excluded if they take/have taken chronically high doses of immunosuppressants or other immune modifying drugs within six months before vaccination, or immunoglobulins or blood products within three months before vaccination, or any investigational product within 30 days before vaccination
* Have a history of influenza infection since previous vaccination
* Women who are pregnant
* Subjects who have an acute or chronic clinically significant disease or an immunosuppressive/deficient condition, or have contra-indications to influenza vaccination

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2006-10; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Evaluation of the safety and reactogenicity of repeated vaccination with adjuvanted influenza vaccine during the 21 days following administration of the vaccine

SECONDARY OUTCOMES:
Evaluation of the humoral immune response and cell-mediated immune response 21 days after revaccination with candidate vaccine

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 104887 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 104887 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 104887 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 104887 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 104887 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 104887 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register